CLINICAL TRIAL: NCT03069612
Title: Evaluating Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Cannabis Dependence and Working Memory in Patients With Early Psychosis
Brief Title: rTMS Treatment for Cannabis Use Disorders in Psychosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Mera Barr, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215/2016
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Cannabis Use Disorder; Psychosis
Keywords: repetitive transcranial magnetic stimulation; working memory; gamma oscillations; dorsolateral prefrontal cortex
MeSH Terms: conditions — Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS Active Group (Experimental): Repetitive transcranial magnetic stimulation (rTMS) will be administered bilaterally to the dorsolateral prefrontal cortex (DLPFC) at 20 Hz, 90% RMT in 25 trains.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- rTMS Sham Group (Sham Comparator): Repetitive transcranial magnetic stimulation (rTMS) will be administered bilaterally to the dorsolateral prefrontal cortex (DLPFC) at 20 Hz, 90% RMT in 25 trains with a sham coil.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS administered bilaterally to the DLPFC at 20 Hz, 90% RMT, 25 trains

SUMMARY:
Cannabis use during adolescence represents a significant risk factor for the development of psychosis including schizophrenia. Moreover, cannabis is the most commonly used drug among patients with an existing psychotic disorder. An estimated 25% of patients with psychosis reportedly meet the criteria of a cannabis use disorder particularly among younger patients experiencing their first episode. Cannabis use significantly exacerbates symptomatology resulting in an increased duration of the first hospitalization visit, number of hospital readmissions, and overall reduced functional outcome. Discovering novel strategies to treat the underlying pathophysiology of cannabis dependence early in the disorder may translate into improved functional outcome. Working memory deficits have been shown to predict relapse in the first-year of psychosis and is modulated with cannabis use. Repetitive transcranial magnetic stimulation (rTMS) targeted to the dorsolateral prefrontal cortex (DLPFC) has shown tremendous promise for the treatment of both tobacco dependence and working memory impairment in patients with psychosis possibly through the modulation of gamma (30-50 Hz) oscillations. The proposed study will therefore evaluate the effect of rTMS on abstinence, working memory performance, and gamma oscillations through a randomized, double-blind, placebo-controlled 28-day longitudinal abstinence study design in patients with early psychosis. It will further explore if baseline performance and gamma oscillations predict abstinence in response to rTMS. It is hypothesized that active compared to sham rTMS will improve abstinence rates and improve working memory performance through the modulation of gamma oscillations.

DETAILED DESCRIPTION:
This a randomized, double-blind placebo-controlled, longitudinal 28-Day abstinence study design. Patients with psychosis will be randomized (1:1) to receive either active or sham stimulation that will be administered three times per week for 4 weeks (28 days) for a total of 12 treatments. Urine will be collected three times per week prior to the rTMS treatment. Cognition including the N-Back task and MATRICS cognitive battery will be administered on Day 0, Day 28, and Day 42 to determine the effect of rTMS on cognition compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-35
* Meet Diagnostic and Statistical Manual for Mental Disorders (DSM)-5 diagnostic criteria for a cannabis use disorder with physiological evidence of dependence; plus one of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, bipolar I disorder, major depressive disorder with psychotic features, cannabis-induced psychosis, or psychosis not otherwise specified
* Full scale IQ ≥ 80 determined through the Wechler Test for Adult Reading (WTAR)
* Daily cigarette smoker of ≥ 5 cigarettes per day

Exclusion Criteria:

* DSM-5 diagnoses of alcohol, substance or poly-use substance use disorder in the past 6 months (other than cannabis/caffeine or nicotine)
* Currently active suicidal ideation or self-harm (suicidal or non-suicidal)
* Head injury resulting in loss of consciousness and hospitalization
* Major neurological or medical illness including seizure disorder or syncope
* Metallic implants
* History of rTMS treatment
* Pregnancy

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Cannabis Abstinence | Change of COOH and creatinine concentrations.from baseline to Day 28.
  Gas chromatography/mass spectrometry (GC/MS) analysis to obtain quantitative THC-COOH and creatinine concentrations.

SECONDARY OUTCOMES:
Working Memory Performance | Baseline, trial endpoint (Day 28) and at follow up (Day 56) for a total of 3 times.
  Working memory task will measure accuracy and reaction time.
Gamma Oscillations | Baseline, trial endpoint (Day 28) and at follow up (Day 56) for a total of 3 times.
  Oscillatory activity will be measured through EEG while performing the working memory task.

CONTACTS AND LOCATIONS:
Overall Officials: Mera S Barr, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating CentreStudy Data/Documents: — http://www.camh.net/research